CLINICAL TRIAL: NCT06101095
Title: A Phase 4, Randomized, Multicenter, Double-blind, Parallel-group, 24 Weeks, Placebo-controlled Study Followed by 104 Weeks Open-label to Assess Dupilumab Efficacy on Esophageal Function and Remodeling in Adult Participants With Eosinophilic Esophagitis (EoE)
Brief Title: A Study Assessing Esophageal Function and Remodeling With Dupilumab Compared With Placebo for 24 Weeks Followed by 104 Weeks Open Label in Adult Participants With EoE (REMOdeling With Dupilumab in Eosinophilic Esophagitis Long-term Trial)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LPS17558; U1111-1280-5266 (Registry Identifier: ICTRP); 2022-502491-23 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Eosinophilic Oesophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Subcutaneous injection (SC) as per protocol
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): SC injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — Subcutaneous injection (SC) as per protocol
  Arms: Dupilumab
Drug: Placebo — SC injection as per protocol
  Arms: Placebo

SUMMARY:
This is parallel, Phase 4 study which consists of a 24 week (0.5 years) randomized, double blind, placebo controlled, 2-arm treatment period followed by an open label segment of 104 weeks (2 years) for a total of 128 weeks (2.5 years) to evaluate the effect of dupilumab treatment on esophageal function, and remodeling in adults with eosinophilic esophagitis.

Duration of study period (per participant)

* Screening period: Up to 12 weeks before Week 0
* Randomized double-blind period: 24 weeks
* Open label period: 104 weeks
* Post Investigational Medicinal Product (IMP) intervention follow-up period: up to 12 weeks or until the participants switch to commercialized dupilumab, whatever comes first.

There will be ten (10) site visits, and five (5) direct-to-participant IMP delivery visits (except if prohibited by local regulatory authorities or if participant is not willing. In this case, IMP will be dispensed at the study site).

DETAILED DESCRIPTION:
The duration per participant will be up to 152 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A documented diagnosis of EoE by endoscopic biopsy.
* Baseline endoscopic biopsies with a demonstration on central reading of intraepithelial eosinophilic infiltration.
* History (by participant report) of an average of at least 2 episodes of dysphagia (with intake of solids) per week in the 4 weeks prior to screening.
* Body weight ≥40 kg.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Other causes of esophageal eosinophilia or the following conditions: hypereosinophilic syndrome or eosinophilic granulomatosis with polyangiitis (Churg Strauss syndrome).
* Active Helicobacter pylori infection.
* History of achalasia, Crohn's disease, ulcerative colitis, celiac disease, and prior esophageal surgery.
* Any esophageal stricture unable to be passed with a standard, diagnostic, 9 to10 mm upper endoscope or any critical esophageal stricture that requires dilation at screening.
* History of bleeding disorders or esophageal varices.
* Treatment with swallowed topical corticosteroids within 8 weeks prior to baseline.
* Initiation or change of a food elimination diet regimen or reintroduction of a previously eliminated food group in the 6 weeks prior to screening.
* Participation in prior dupilumab clinical study or participants currently treated or have been treated with commercially available dupilumab or contraindicated to dupilumab per local labelling.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in esophageal distensibility plateau as measured by Functional Lumen Imaging Probe (EndoFLIP) | From baseline to Week 24
  Distensibility plateau provides an assessment of esophageal function. An increase in distensibility plateau indicates an improvement in esophageal function and a decrease in distensibility plateau indicates a worsening of esophageal function.

SECONDARY OUTCOMES:
Percent change from baseline in esophageal distensibility plateau as measured by Functional Lumen Imaging Probe | From baseline up to Week 24
  Distensibility plateau provides an assessment of esophageal function. An increase in distensibility plateau indicates an improvement in esophageal function and a decrease in distensibility plateau indicates a worsening of esophageal function.
Absolute change from baseline in esophageal distensibility plateau as measured by Functional Lumen Imaging Probe | From baseline up to Week128
  Distensibility plateau provides an assessment of esophageal function. An increase in distensibility plateau indicates an improvement in esophageal function and a decrease in distensibility plateau indicates a worsening of esophageal function.
Percent change from baseline in esophageal distensibility plateau as measured by Functional Lumen Imaging Probe | From Baseline up to Week 128
  Distensibility plateau provides an assessment of esophageal function. An increase in distensibility plateau indicates an improvement in esophageal function and a decrease in distensibility plateau indicates a worsening of esophageal function.
Change from baseline in eosinophilic esophagitis-endoscopic reference score (EoE-EREFS) | From baseline up to Week 128
  EoE-EREFS, a scoring system for inflammatory and remodeling features of disease. The overall total score ranges from 0 to 18 with higher number indicating worse disease.
Change from baseline in eosinophilic esophagitis (EoE-HSS) Grade | From Baseline up to Week 128
  Severity (grade) and extent (stage) of esophageal abnormalities are scored using a 4-point scale (0 normal; 3 maximum change). Higher score indicates greater severity and extent of histological abnormalities.
Change from baseline in EoE-HSS Stage | From Baseline up to Week 128
  Severity (grade) and extent (stage) of esophageal abnormalities are scored using a 4-point scale (0 normal; 3 maximum change). Higher score indicates greater severity and extent of histological abnormalities.
Proportion of participants who achieved peak Esophageal Intraepithelial Eosinophil Count of ≤6 eosinophils/high power field (Eos/HPF) | At Weeks 24, 76 and 128
  Esophageal intraepithelial eosinophil count obtained by esophageal endoscopy with biopsies (all 3 esophageal regions: proximal, mid, and distal).
Proportion of participants who achieved peak Esophageal Intraepithelial Eosinophil Count of ≤15 Eos/HPF | At Weeks 24, 76 and 128
  Esophageal intraepithelial eosinophil count obtained by esophageal endoscopy with biopsies (all 3 esophageal regions: proximal, mid, and distal).
Change from baseline in normalized enrichment score (NES) for EoE diagnostic panel (EDP) transcriptome signature | From baseline up to Week 128 (EOT)
  NES reflects the degree to which the activity level of a set of disease transcripts is overrepresented at the extremes (top or bottom) of the entire ranked list of transcripts within a sample and is normalized by accounting for the number of transcripts in the set. An NES of 0 indicates no change from baseline, a negative score reflects a reduction in the disease score (more like normal) and a positive score reflects worsening (more active disease).
Change from baseline in normalized enrichment score (NES) for type 2 inflammation transcriptome signature | From Baseline up to Week 128 (EOT)
  NES reflects the degree to which the activity level of a set of disease transcripts is overrepresented at the extremes (top or bottom) of the entire ranked list of transcripts within a sample and is normalized by accounting for the number of transcripts in the set. An NES of 0 indicates no change from baseline, a negative score reflects a reduction in the disease score (more like normal) and a positive score reflects worsening (more active disease).
Incidence of treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs) | From the first IMP administration up to end of post treatment follow up period (week139)
Incidence of adverse events of special interest (AESIs) | From the first IMP administration up to end of post treatment follow up period (week139)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (30):
- United States (15):
  - United Gastroenterologists - Murrieta- Site Number : 8400001, Murrieta, California
  - University of California San Francisco - Parnassus Heights- Site Number : 8400020, San Francisco, California
  - Borland Groover Clinic- Site Number : 8400016, Jacksonville, Florida
  - Treasure Valley Medical Research- Site Number : 8400018, Boise, Idaho
  - Northwestern University- Site Number : 8400003, Chicago, Illinois
  - GI Alliance - Glenview- Site Number : 8400012, Glenview, Illinois
  - Illinois Gastroenterology Group- Site Number : 8400004, Gurnee, Illinois
  - University of Iowa- Site Number : 8400006, Iowa City, Iowa
  - University of Massachusetts Chan Medical School- Site Number : 8400019, Worcester, Massachusetts
  - Mayo Clinic Hospital Rochester- Site Number : 8400008, Rochester, Minnesota
  - University of North Carolina at Chapel Hill- Site Number : 8400007, Chapel Hill, North Carolina
  - Cleveland Clinic - Cleveland- Site Number : 8400009, Cleveland, Ohio
  - Penn Medicine: University of Pennsylvania Health System- Site Number : 8400010, Philadelphia, Pennsylvania
  - Private Practice - Dr. Martin Yudovich- Site Number : 8400015, Houston, Texas
  - GI Alliance - Mansfield- Site Number : 8400017, Mansfield, Texas
- Brazil (5):
  - Itaigara Memorial - Hospital Dia- Site Number : 0760005, Salvador, Estado de Bahia
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760006, Porto Alegre, Rio Grande do Sul
  - Clínica Loema - Unidade I- Site Number : 0760007, Campinas, São Paulo
  - Clinica de Alergia Martti Antila- Site Number : 0760001, Sorocaba, São Paulo
  - Hospital Alemao Oswaldo Cruz - São Paulo- Site Number : 0760003, São Paulo
- Canada (3):
  - Investigational Site Number : 1240006, Vancouver, British Columbia
  - Investigational Site Number : 1240004, Vancouver, British Columbia
  - Investigational Site Number : 1240002, Montreal, Quebec
- Israel (5):
  - Investigational Site Number : 3760006, Haifa
  - Investigational Site Number : 3760002, Haifa
  - Investigational Site Number : 3760005, Jerusalem
  - Investigational Site Number : 3760004, Jerusalem
  - Investigational Site Number : 3760003, Tel Aviv
- Switzerland (2):
  - Investigational Site Number : 7560001, Wetzikon
  - Investigational Site Number : 7560002, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Dellon ES, Savarino EV, Zaghloul S, Angello JT, Zhang M, Raphael BP, Radwan A, Bredenoord AJ. Study design of the phase IV, randomized, placebo-controlled REMOdeling with Dupilumab in Eosinophilic esophagitis Long-term (REMODEL) trial. Therap Adv Gastroenterol. 2025 Oct 9;18:17562848251383782. doi: 10.1177/17562848251383782. eCollection 2025. PMID 41084592
- See also: LPS17558 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25510&tenant=MT_SNY_9011